CLINICAL TRIAL: NCT05510115
Title: Feasibility of Study of Empagliflozin in Patients With Autosomal Dominant Polycystic Kidney Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-0616; 1R01DK131755-01A1 (NIH)
Record Dates: First submitted 2022-08-11; First posted 2022-08-22 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Polycystic Kidney, Autosomal Dominant
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Empagliflozin
  Interventions: Drug: Empagliflozin
- Placebo comparator (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin: The chemical name of empagliflozin is D-Glucitol,1,5-anhydro-1-C-[4-chloro-3-[[4-[[(3S)-tetrahydro-3furanyl]oxy]phenyl]methyl]phenyl]-, (1S). Empagliflozin is a white to yellowish, non-hygroscopic powder. It is very slightly soluble in water, sparingly soluble in methanol, slightly soluble in ethanol and acetonitrile; soluble in 50% acetonitrile/water; and practically insoluble in toluene. Empagliflozin power will be added in white and bovine origin gelatin capsules. Each capsule of empagliflozin will contain 10 mg or 25 mg of empagliflozin (free base) and the following inactive ingredients: microcrystalline cellulose magnesium, stearate, dicalcium phosphate, and silicone dioxide.
  Arms: Experimental
Drug: Placebo — Placebo capsules will be matched in size and color to empagliflozin capsules. Each placebo capsule will contain the following inactive ingredients: microcrystalline cellulose magnesium, stearate, dicalcium phosphate, and silicone dioxide.
  Arms: Placebo comparator

SUMMARY:
The investigator proposes a pilot randomized clinical trial to determine the safety and tolerability of empagliflozin in ADPKD patients. To achieve this, the investigator will conduct a 12-month parallel-group, randomized, double-blind, placebo-controlled trial in 50 ADPKD patients with an eGFR 30-90 mL/min/1.73m2.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is characterized by development and continued growth of numerous fluid-filled kidney cysts that result in ultimate loss of kidney function in the majority of individuals. ADPKD manifestations are not limited to the kidney. It is well established that arterial stiffness, an important predictor of future cardiovascular events and mortality, is present early in the course of ADPKD. Sodium-glucose cotransporters-2 inhibitors (SGLT2i) have a track record of tolerability and safety in patients with diabetic and non-diabetic kidney disease. Studies of SGLT2i have been extremely encouraging and the expectation is that these treatments will become standard of care for diabetic and non-diabetic kidney disease; however, the mechanism of action is not fully understood and seems non-specific with regards to disease etiology. The potential benefit of SGLT2i has not been examined in ADPKD, as major trials of SGLT2i in non-diabetic chronic kidney disease (CKD) have excluded patients with ADPKD. It is also important to note the potential benefits of SGLT2i outside of delaying loss of kidney function, as these class of drugs have been shown to provide a mortality benefit for patients across the CKD spectrum. Thus, novel interventions to slow kidney disease progression and reduce vascular morbidity within ADPKD population are of clinical importance.

Limited data suggests SGLT2i may stimulate vasopressin and vasopressin receptor expression by causing glucosuria, natriuresis, and glucose osmotic diuresis, at least in patients and animal models without ADPKD. Vasopressin is known to stimulate cyst growth in ADPKD and promote disease progression. SGLT2i have been studied in animal models of ADPKD, with conflicting data. Some studies in rodent ADPKD models treated with SGLT2i failed to show a significant reduction in cyst growth. However, because of SGLT2i's beneficial effects on kidney function, vascular function, and mortality in non-ADPKD patients with CKD, further investigations of SGLT2i in patients with ADPKD are needed.

Primary Outcome Measure (Aim1): Safety will be assessed by laboratory testing and recording of adverse events. Tolerability will be assessed by subject drop-out rate due to adverse events and the proportion tolerating the maximal dose of study drug. Adherence to the intervention will be assessed by counting the returned number of tablets during check-in visits. Subjects will have check-in visits every 2 weeks the 1st month, monthly on month 2 and 3 and then every 3 months until the end of the study. Subjects will discuss issues with tolerability or treatment-emergent adverse events with a member of the clinical staff who is blinded to treatment status.

Secondary (Exploratory) Outcome Measures (Aim 2): (a) Height-adjusted total kidney volume will be examined by magnetic resonance imaging, at baseline, 3 months and 12 months after treatment with empagliflozin or placebo; (b) Aortic stiffness will be evaluated as aortic pulse wave velocity, at baseline, 3 months and 12 months after treatment with empagliflozin or placebo; (c) Plasma copeptin levels and urinary kidney injury molecule-1 will be measured at baseline, 3 months and 12 months after treatment with empagliflozin or placebo; and (d) Patient related outcomes will be measured using the ADPKD Impact Scale (ADPKD-IS) at baseline, 3 months and 12 months after treatment with empagliflozin or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Autosomal Dominant Polycystic Kidney Disease (ADPKD) as defined by modified Pei-Ravine Criteria;
* Age 18-55 yrs;
* Estimated Glomerular Filtration Rate (eGFR) 30-90 ml/min/1.73m2;
* Mayo imaging-based risk classification 1C, 1D, or 1E;
* Stable renal function over prior 3 months.

Exclusion Criteria:

* Known diabetes mellitus;
* Fasting Glucose >120 mg/dL;
* HbA1C≥6.5%;
* Seated systolic blood pressure <100 mm Hg;
* Seated systolic blood pressure >160 mm Hg;
* Known heart failure with reduced ejection fraction (HFrEF);
* Current use of loop diuretic;
* Current use of tolvaptan or other V2 receptor antagonist;
* Current urinary tract or urogenital infection;
* Pregnant or lactating;
* Vascular claudication, lower extremity skin infection or ulcers;
* Contraindication to magnetic resonance imaging (e.g., severe claustrophobia, implanted ferromagnetic device).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 12 months
  Safety will be assessed by recording of adverse events.
Subject Drop Out Rate | 12 months
  Tolerability will be assessed by subject drop-out rate due to adverse events and maximal tolerated dose.
Returned Number of Tablets | 12 months
  Adherence to the intervention will be assessed by counting the returned number of tablets during check-in visits.

SECONDARY OUTCOMES:
Height-Adjusted Total kidney volume | Baseline, check-in visit (3 months), post-testing (12-months)
  To assess kidney growth, we will measure change in height-adjusted total kidney volume by magnetic resonance imaging at baseline, 3 months and 12 months.
Aortic Pulse Wave Velocity (aPWV) | Baseline, check-in visit (3 months), post-testing (12 months)
  A transcutaneous custom tonometer (SphygmoCor XCEL PWA and PWV System; Atcor Medical Inc, Naperville IL) will be positioned at the carotid and femoral arteries and aPWV will be calculated as the distance between recording sites/time between the foot of the carotid and femoral arterial waveforms. Data will be expressed as cm/s.
Mechanistic Biomarkers | Baseline, check-in visit (3 months), post-testing (12 months)
  Venous blood samples will be analyzed for the following circulating mechanistic biomarker: Plasma copeptin.
  Urine samples will be analyzed for the following mechanistic biomarker:
  Kidney Injury Molecule -1 (KIM-1).
Patient Related Outcomes | 12 months
  The ADPKD Impact Scale (ADPKD-IS) includes 18 items representing 3 distinct domains (physical function, fatigue, and emotional function

CONTACTS AND LOCATIONS:
Overall Officials: Michel B Chonchol, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Coloardo Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
All NIH applicable guidelines regarding data sharing will be followed. At the conclusion of the study, data that is coded with a number will be made available to qualified individuals within the scientific community who apply for data use. The results and outcomes of the studies will be made generally available by publication with journal articles submitted to PubMed Central in compliance with NIH access guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: NIH applicable guidelines regarding data sharing will be followed.
Access Criteria: NIH applicable guidelines regarding data sharing will be followed.

REFERENCES:
- [Derived] Eswarappa M, Madden E, Shlipak MG, Cui X, Mrug M, Estrella MM, Park M. Sodium-Glucose Cotransporter-2 Inhibitor Therapy and Longitudinal Changes in Kidney Function among Veterans with Autosomal Dominant Polycystic Kidney Disease. Clin J Am Soc Nephrol. 2025 May 16;20(7):940-949. doi: 10.2215/CJN.0000000725. PMID 40377984
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Hogan MC, Simmons K, Ullman L Jr, Gondal M, Dahl NK. Beyond Loss of Kidney Function: Patient Care in Autosomal Dominant Polycystic Kidney Disease. Kidney360. 2023 Dec 1;4(12):1806-1815. doi: 10.34067/KID.0000000000000296. Epub 2023 Nov 27. PMID 38010035